CLINICAL TRIAL: NCT05835232
Title: Sleep Disorders, Mental Health and Quality of Life in a Court of HIV+ Patients
Brief Title: Sleep Disorders and Psychophysical Well-being in HIV+ Patients
Acronym: DISOMETA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5250
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Each participant completed an anonymous 62-item online survey.

SUMMARY:
The primary goal of this observational study is to investigate sleep quality in patients living with HIV+. The secondary objective is to measure the influence of sleep quality on indicators of mental health (anxiety, depression and stress) and quality of life.

The main questions it aims to answer are:

* Measuring the effects of poor sleep quality on mental and physical health in HIV+ patients.
* Monitor the sleep pattern in the HIV+ population.

Participants will fill out an online cross-sectional survey.

The online questionnaire survey will collect:

* sociodemographic and clinical data related to HIV infection,
* sleep quality,
* mental health,
* quality of life.

ELIGIBILITY:
Inclusion Criteria:

* HIV diagnosis.
* Being treated at the Infectious Diseases Outpatient Clinic of Policlinico Gemelli in Rome.
* Ongoing antiretroviral therapy.
* Age > 18 years.
* Native Italian speaker.
* Informed consent to participate in the study

Exclusion Criteria:

* Absence of an HIV diagnosis.
* Not being treated at the Infectious Diseases Outpatient Clinic of Policlinico Gemelli in Rome.
* Absence of ongoing antiretroviral therapy.
* Age > 18 years.
* Not being a native Italian speaker.
* Refusal to sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expect the majority of the HIV patient population to be male, between the ages of 40 and 65 and with a high school diploma. We expect a virologically suppressed HIV population with good adherence to antiretroviral therapy. We expect poor sleep quality and low quality of life and high symptoms of depression, anxiety and stress.
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | 1 year
  It will investigate with the Italian version of the Pittsburgh Sleep Quality Index (PSQI) the quality of sleep in HIV+ patients by assessing the reported subjective quality, latency, duration, efficiency, degree of disturbed sleep, use of sleep medications, and how much sleep-related problems affect daily routines.

SECONDARY OUTCOMES:
Influence of sleep quality on mental health | 1 year
  Mental health will be investigated using the Depression Anxiety Stress Scale (DASS) 21, a self-assessment instrument containing 21 useful items to investigate three constructs: depression, anxiety and stress. Each construct constitutes a specific subscale, consisting of 7 items. Each item corresponds to a statement, referring to the past week.
Influence of sleep quality on quality of life | 1 year
  Quality of life will be investigated using the 12-item Short-Form Health Survey (SF-12). The SF-12 investigates quality of life with 12 items: 6 items are concerned with physical health (physical functioning, physical plane limitations, physical pain, general health) and 6 items are concerned with mental health (emotional plane limitations, fatigue or lack of energy, social functioning, emotional well-being).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No